CLINICAL TRIAL: NCT03272321
Title: Influence of Oxytocin on Neurophysiological Responses to Direct and Averted Gaze
Brief Title: Influence of Oxytocin on Neurophysiological Responses to Live Faces
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Kaat Alaerts, Prof. Dr. Kaat Alaerts, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SingleOT_EEG-SC_S56327
Record Dates: First submitted 2017-08-25; First posted 2017-09-05 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Oxytocin
Keywords: biomedical intervention; oxytocin; EEG; skin conductance response; heart rate; gaze direction; eye contact
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Syntocinon nasal spray (40 IU/ml; oxytocin, product code RVG 03716); single intranasal dose of 24 international units (IU; 3 puffs of 4 IU per nostril)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): saline natriumchloride solution nasal spray; single intranasal dose (3 puffs per nostril)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Syntocinon nasal spray
  Other Names: syntocinon
  Arms: Oxytocin
Drug: Placebo — Placebo nasal spray
  Arms: Placebo

SUMMARY:
Previous research has indicated that direct eye gaze compared to averted gaze, elicits a higher skin conductance response (SCR), and a more pronounced left frontal cortex activity than right frontal cortex activity (resulting in positive asymmetry scores). On a behavioral level, participants tend to look shorter at live faces with a direct gaze as compared to averted gaze (Akechi et al., 2013). Further, subjective evaluations showed that a direct gaze is rated more arousing and less pleasant than an averted gaze (Akechi et al., 2013; Hietanen, Leppänen, Peltola, Linna-aho, & Ruuhiala, 2008).

Importantly, oxytocin administration increases the number of fixations and to looking time towards the eye region during live social interaction. Further, oxytocin has been shown to influence SCR and heart rate variability. Therefore, it is conceivable that oxytocin will not only influence the gaze duration of the participant, but also the physiological and neurological responses elicited by direct eye gaze.

In this study, the investigators will investigate whether oxytocin modulates the behavioural (eye gaze and subjective ratings), neurological (EEG) and physiological (skin conductance, heart rate and respiration) responses elicited by direct gaze.

DETAILED DESCRIPTION:
Previous research has indicated that direct eye gaze compared to averted gaze, elicits a higher skin conductance response (SCR), and a more pronounced left frontal cortex activity than right frontal cortex activity (resulting in positive asymmetry scores). On a behavioral level, participants tend to look shorter at live faces with a direct gaze as compared to averted gaze (Akechi et al., 2013). Further, subjective evaluations showed that a direct gaze is rated more arousing and less pleasant than an averted gaze (Akechi et al., 2013; Hietanen, Leppänen, Peltola, Linna-aho, & Ruuhiala, 2008).

Importantly, oxytocin administration increases the number of fixations and to looking time towards the eye region during live social interaction. Further, oxytocin has been shown to influence SCR and heart rate variability. Therefore, it is conceivable that oxytocin will not only influence the gaze duration of the participant, but also the physiological and neurological responses elicited by direct eye gaze.

In this randomized, placebo controlled, double blinded study, the investigators will investigate whether oxytocin modulates the behavioral and neurophysiological responses elicited by direct gaze. In order to do so, the investigators will measure behavioural (eye gaze and subjective feelings), physiological (skin conductance, blood volume pulse, and respiration) and neurological (EEG) responses during presentations of a live person's face with direct gaze and closed eyes, before and after oxytocin or placebo administration.

The investigators hypotheses that oxytocin attenuates the heightened SCR and pronounced EEG asymmetry during direct gaze. Further, they expect that oxytocin increases the number of fixations and duration of those fixations towards the eye region. Exploratory, the investigators will also investigate whether oxytocin administration influences respiration and the subjective reports on experience of live eye contact. Lastly (and also exploratory), they will explore whether certain personality traits (as measured by SAAM (state adult attachment measure) and SRS (social responsiveness scale)) influence the modulatory effect of oxytocin on neurological and behavioural responses.

Note that this study is part of a larger study in which the investigators also register several neurophysiological responses (blood volume pulse, respiration, heart rate, EEG, skin conductance) during rest before and after oxytocin or placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* male
* age between 18 and 35
* Normal or adjusted-to-normal vision (with lenses only)
* Dutch as mother tongue

Exclusion Criteria:

* not right-handed
* female
* age below 18 or above 35
* Need to wear glasses
* Dutch not as mother tongue

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Change in EEG asymmetry after oxytocin administration | Average over several trials, baseline and 40 min after oxytocin or placebo administration
  The influence of oxytocin administration on EEG asymmetry
Change in skin conductance (type of electrodermal activity) response after oxytocin administration | Average over several trials, baseline and 40 min after oxytocin or placebo administration
  The influence of oxytocin administration on skin conductance response

SECONDARY OUTCOMES:
Change in duration of fixations to face regions after oxytocin administration | Assesment over several trials, baseline and 40 min after oxytocin or placebo administration
  The influence of oxytocin administration on gaze behavior (duration of fixation to upper and lower face regions)
Change in number of fixations to face regions after oxytocin administration | Assesment over several trials, baseline and 40 min after oxytocin or placebo administration
  The influence of oxytocin administration on gaze behavior (number of fixation to upper and lower face regions)

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Alaerts, PhD, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium